CLINICAL TRIAL: NCT00615758
Title: ERLOTINIB, A TYROSINE KINASE INHIBITOR OF EPIDERMAL GROWTH FACTOR RECEPTOR (EGFR) AS FIRST LINE TREATMENT, IN PATIENTS WITH LOCALLY ADVANCED/METASTATIC NON SMALL CELL LUNG CANCER (NSCLC). A PHASE II STUDY
Brief Title: Erlotinib as 1st Line Treatment in NSCLC Stage IIIB/IV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: V.Georgoulias, Hellenic Oncology Research Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/06.03
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Erlotinib; Biological therapy; Tyrosin Kinase Inhibitor therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Tarceva
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib at the dose of 150 mg orally once a day continually until progression
  Other Names: Tarceva

SUMMARY:
To evaluate the efficacy and toxicity of erlotinib as first line treatment in patients with locally advanced/metastatic (stages IIIB/IV) NSCLC, with clinical predictors of response to tyrosine kinase inhibitors (erlotinib, gefitinib), such as female gender, never-smoking status and adenocarcinoma histology. Furthermore, erlotinib-sensitivity will be correlated with the presence of EGFR mutations in exons 18, 19 and 21, in this population

DETAILED DESCRIPTION:
A randomized, placebo-controlled phase III trial of erlotinib versus placebo, with more than 700 patients demonstrated that therapy with this tyrosine kinase inhibitor (TKI) prolongs survival after first or second line therapy in patients with advanced NSCLC. Statistically significant and clinically relevant differences were observed for overall and progression free survival in favour of erlotinib. Moreover, several clinical factors had been correlated with response to gefitinib or erlotinib, including never smoking status, female gender, Asian ethnicity and adenocarcinoma histology (especially bronchioalveolar carcinoma).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, unresectable locally advanced (stage IIIB with pleural effusion) and/or metastatic (stage IV) NSCLC
* No previous therapy for advanced/metastatic NSCLC is allowed
* age >18 years
* bidimensionally measurable disease
* non-smokers (or ex-smokers with less than 5 pack-years smoking history)
* adenocarcinoma histology
* performance status (WHO) 0-3
* adequate liver (serum bilirubin <1.5 times the upper normal limit (UNL); AST and ALT <2.5 times the UNL in the absence of demonstrable liver metastases, or <5 times the UNL in the presence of liver metastases); adequate renal function (serum creatinine <1.5 times the UNL); and bone marrow (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L) function
* previous radiotherapy, either in the adjuvant setting or for the treatment of metastatic disease is allowed provided that the measurable lesions are outside the radiation fields
* patient able to take oral medication
* tissue sample for tumour mutational analysis is required

Exclusion Criteria:

* serious chronic skin conditions (e.g. psoriasis, eczema) that would preclude study participation
* active infection
* history of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* malnutrition (loss of ≥ 20% of the original body weight)
* performance status: 4
* psychiatric illness or social situation that would preclude study compliance
* pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Overall Survival | 1-year OS
Time to Tumor Progression | 1 year TTP
Quality of life assessment | Assessment every two cycles
Toxicity assesment | Toxicity assessment on each cycles

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete; Athanasios Pallis, MD, Principal Investigator — University Hospital of Crete
Locations (5):
- Greece (5):
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - Sotiria" General Hospital, 2nd Dep of Pulmonary Diseases, Athens
  - "Diabalkaniko" Anticancer Hospital of Thessaloniki, Thessaloniki